CLINICAL TRIAL: NCT04997083
Title: Evaluation of the Treatment Outcome of Cleft Palate Patients Treated With Differential Opening Expander With Slow Protocol and Face Mask
Brief Title: Slow Expansion and Protraction in Cleft Lip and Palate Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Amira Helmy Abdulsattar Eldawy, Principal Investigator, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2-D
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cleft Lip and Palate
Keywords: Cleft lip and palate; Expansion; Slow expansion; Maxillary expander with differential opening (EDO); Protraction; Face mask; Cone beam computed tomography (CBCT)
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cleft lip and palate patients (Experimental): Cleft patients with transverse maxillary constriction and anteroposterior deficiency
  Interventions: Device: Maxillary Expander with Differential Opening (EDO); Device: Petit face mask

INTERVENTIONS:
Device: Maxillary Expander with Differential Opening (EDO) — The EDO is designed with two expansion screws positioned transversely. When more expansion is required between the canines, the anterior screw can be further activated. Both expansion screws can be activated to open in a parallel configuration. Pivoting corner screws allow for different amounts of expansion without significant risk of binding during activation.
Device: Petit face mask — The face mask is anatomical, multi-adjustable, lightweight and an ideal therapeutic alternative for the correction of Class III malocclusion. It consists of forehead cap, chin cap, and cross bar.

SUMMARY:
Evaluate the treatment outcome of slow maxillary expansion protocol on patients with cleft lip and palate, using a differential opening expander and face mask which will be measured and recorded by cone beam computed tomography (CBCT).

DETAILED DESCRIPTION:
Cleft lip and palate are among the most common deformities in children. Cleft patients are usually having orofacial problems as missing or unerupted permanent teeth, alveolar bone defect, speech difficulty. Patients with cleft lip and palate (CLP) commonly have maxillary arch constriction (maxillary hypoplasia) and Class III malocclusions due to deficient of maxillary growth. The upper jaw of patients with cleft palate will be expanded using maxillary Expander with Differential Opening (EDO) which has two screws; one anterior and one posterior. This will be done with slow expansion protocol, which is one 1/4 turn three times weekly. Petit facemask will be used to protract the retracted maxilla. The differences in measurements between before and after treatment will be assessed by cone beam computed tomography (CBCT).

ELIGIBILITY:
Inclusion Criteria:

* All patient age ranges from 8 to 12 years.
* Patients of both sexes.
* Cleft lip and palate patients.
* All the cases showed maxillary arch constriction and deficiency.
* All patients had maxillary permanent first molars.
* Primary lip adhesion and palatal closure.

Exclusion Criteria:

* Patients had received any surgical assisted rapid maxillary expansion or maxillary protraction of fixed orthodontics before.
* Maxillary dentition unsuitable to bond the expander (less than two dental units beside permanent first molar).
* Absent maxillary permanent first molars.
* Uncooperative patients/parents.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Changes in 3 dimensions of skull before and after expansion | Six months
  Full skull Cone Beam Computerized Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Amany M. Diab, PhD, Study Director — Lecturer of Orthodontics Department, Faculty of Dental Medicine for Girls, Al-Azhar University
Locations (1):
- Faculty of dental medicine for girls, Al-Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No
Evaluation of EDO, Slow maxillary expansion and facemask in patients with cleft lip and palate (CLP) using Cone Beam Computed Tomography (CBCT)

REFERENCES:
- [Background] Alves ACM, Janson G, Mcnamara JA Jr, Lauris JRP, Garib DG. Maxillary expander with differential opening vs Hyrax expander: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2020 Jan;157(1):7-18. doi: 10.1016/j.ajodo.2019.07.010. PMID 31901284
- [Background] Massaro C, Garib D, Cevidanes L, Janson G, Yatabe M, Lauris JRP, Ruellas AC. Maxillary dentoskeletal outcomes of the expander with differential opening and the fan-type expander: a randomized controlled trial. Clin Oral Investig. 2021 Sep;25(9):5247-5256. doi: 10.1007/s00784-021-03832-9. Epub 2021 Feb 12. PMID 33580351
- See also: Maxillary dentoskeletal outcomes of the expander with differential opening and the fan-type expander: a randomized controlled trial — https://link.springer.com/article/10.1007/s00784-021-03832-9